CLINICAL TRIAL: NCT04223700
Title: Ultrasound-guided Thoracic Spinal Level Identification Using Rhomboid Muscle as a Reference Landmark
Brief Title: Ultrasound-guided Thoracic Spinal Level Identification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Associate Professor, Seoul National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1911-063-1078
Record Dates: First submitted 2019-12-16; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Thoracic Diseases; Myofascial Pain
Keywords: Ultrasound guided intervention; Rhomboid muscle; Thoracic spine
MeSH Terms: conditions — Thoracic Diseases | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group 1 (Experimental): Ultrasound scanning of the rhomboid muscle
  Interventions: Procedure: Ultrasound imaging & fluoroscopic confirmation

INTERVENTIONS:
Procedure: Ultrasound imaging & fluoroscopic confirmation — The researchers use ultrasound to scan the left and right sides of the paravertebral sagittal imaging to identify trapezius, semispinalis, erector spinae muscle, transverse process and rhomboid muscle. The radiopaque marker is attached respectively to the skin of the inferior margin of the rhomboid muscle on the left and right thoracic spinal spines. Then, as the first step for the scheduled nerve block to the patient, thoracic vertebra level verification using C-arm is performed. At this time, left and right level of the transverse process of thoracic spine marked with the radiopaque marker are confirmed and recorded.

SUMMARY:
Typically, the rhomboid minor muscles rise from the C7-T1 spinous process and run downward to touch the upper inner corner of the scapula, and the rhomboid major muscles rise from the T2-T5 spinous process and run downward to reach the lower middle inner corner of the scapula. In anatomical research articles, it has been reported that the rhomboid muscle's anatomical variations are rare. Considering the characteristics of these rhomboid muscles, the investigators planned a study on the utility of rhomboid muscles as a landmark for identifying thoracic spine levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic nerve root block due to herpes zoster, postherpetic neuralgia, complex regional pain syndrome, post traumatic pain syndrome, or compression fracture of vertebra.

Exclusion Criteria:

1. Previous T-spine surgery
2. Patient refusal
3. Coagulopathy
4. Generalized infection or localized infection at injection site
5. Anatomical abnormality of T-spine
6. Allergic reaction to local anesthetics

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-13 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Ultrasound-guided Thoracic Spinal Level | during the procedure
  Thoracic vertebra level of radiopaque marker labeled on the rhomboid muscle inferior margin on C-arm

SECONDARY OUTCOMES:
1. Changes in marker position when raised the arm above the head and in a relaxed position | during the procedure
2. Rhomboid muscle variation | during the procedure
  The presence of rhomboid muscle fusion
3. Visibility grade of muscle fascia using Ultrasound (I - IV) | during the procedure
  A. Grade I: Definitely visible B. Grade II: Somewhat visible C. Grade III: Barely visible D. Grade IV: Not visible
4. Depth: The distance from the skin where the marker is attached to the transverse process of thoracic spine | during the procedure
5. Difference between left and right sides | during the procedure
  The distance between left and right inferior thoracic spine attachment site of rhomboid muscle

REFERENCES:
- [Derived] Jung H, Bae J, Kim J, Yoo Y, Lee HJ, Rho H, Han AH, Moon JY. Can the Rhomboid Major Muscle Be Used to Identify the Thoracic Spinal Segment on Ultrasonography? A Prospective Observational Study. Pain Med. 2022 Sep 30;23(10):1670-1678. doi: 10.1093/pm/pnac043. PMID 35289904